CLINICAL TRIAL: NCT04306874
Title: High-Protein Oral Nutritional Supplementation in Patients Undergoing Pancreaticoduodenectomy
Brief Title: Whipple Protein Study
Acronym: WPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 19D.669; JT 14375 (Other: JeffTrial Number)
Record Dates: First submitted 2019-12-06; First posted 2020-03-13 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Pancreatic Cancer; Malnutrition
Keywords: pancreaticoduodenectomy; surgery; nutrition; protein
MeSH Terms: conditions — Pancreatic Neoplasms; Malnutrition

STUDY DESIGN:
Intervention Model Description: Parallel, non-blinded, randomized controlled two-arm trial: supplement vs. placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Protein Supplement (Experimental): 60 g total protein per day, administered via twice daily ensure max protein shakes
  Interventions: Dietary Supplement: Ensure Max Protein
- Control (No Intervention): No intervention on diet; routine dietary practice

INTERVENTIONS:
Dietary Supplement: Ensure Max Protein — Liquid shake with 30 g protein per serving
  Arms: High Protein Supplement

SUMMARY:
Study investigators aim to assess the effect of providing high-protein nutritional supplementation before and after surgery

DETAILED DESCRIPTION:
Pancreaticoduodenectomy (PD) is a complex and morbid operation that is associated with many potential complications. Many people undergoing PD are malnourished due to their underlying medical condition or difficulties eating in the face of abdominal pain or obstruction from pancreatic disease. This study aims to assess the effect of high-protein dietary supplementation in improving perioperative nutrition and decreasing complications. We will randomize PD patients to an experimental arm in which they take a nutritional, high-protein supplement for 2 weeks before and after surgery, or to a control arm, where they will take a standard postoperative diet without supplementation. Outcomes and nutritional parameters will be examined after they complete the supplements.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing pancreaticoduodenectomy
* Patients aged 18 years and older
* Patients able to provide written informed consent
* Patients able to understand and comply with study guidelines
* Patients able to tolerate oral intake
* Patients who are malnourished or at risk of malnutrition as defined by a score less than 12 on the Mini-Nutritional Assessment

Exclusion Criteria:

* Patients with a milk protein allergy
* Patients with a vegan diet
* Patients dependent on artificial enteral feeding
* Patients with end-stage renal disease undergoing dialysis
* Patients who are pregnant
* Patients with ongoing eating disorder or condition precluding oral intake
* Patients who are scheduled for pancreaticoduodenectomy but are unable to receive this surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-08-20 (Actual); Primary Completion 2022-05-10 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
Complications | 30 days
  All complications within 30 days of surgery

SECONDARY OUTCOMES:
Overall Survival | 6 months
  Overall survival time since surgery
Prealbumin level | 30 days
  Serum prealbumin level (normal 15-36 mg/dL). Lower levels indicate acute malnutrition.

CONTACTS AND LOCATIONS:
Overall Officials: Harish Lavu, MD, Principal Investigator — Associate Professor
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided